CLINICAL TRIAL: NCT01478464
Title: Danish: Integreret Motion på Arbejdspladsen (IRMA) English: Implementation of Exercise at the Workplace
Brief Title: Effect of Massage on Hamstring Muscle Soreness
Acronym: IRMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre for the Working Environment, Denmark (Other Government)
Responsible Party: Principal Investigator, Lars L. Andersen, Principal Investigator, National Research Centre for the Working Environment, Denmark
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: IRMA03
Record Dates: First submitted 2011-11-18; First posted 2011-11-23 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Musculoskeletal Disorders
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Control group, does not receive any intervention
- Massage group (Experimental): Massage will be performed on the left or right hamstring muscle (randomized) for ten minutes with a massage roller. The contralateral leg will not be massaged, but serve as a non-massaged control leg to assess possible cross-over effects from the massaged leg
  Interventions: Other: Massage

INTERVENTIONS:
Other: Massage — The hamstring muscle will be massaged with a "massage roller" for ten minutes.
  Arms: Massage group

SUMMARY:
Delayed onset muscular soreness peaks in 24-48 hours after unaccustomed strenuous physical exercise. Therapists often provide manual massage with the hands to acutely relief the soreness. Alternatives to manual hand massage can be useful for therapists. Here the investigators examine the acute effect of a "massage roller" on DOMS in the hamstring muscles

ELIGIBILITY:
Inclusion Criteria:

* working age adults

Exclusion Criteria:

* blood pressure above 160/100
* disease of the cervical spine

Ages: 18 Years to 67 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Perceived soreness on a scale of 0-10 | change from before to after massage (average of 0, 10, 30 and 60 min after)
  0: no soreness 10: worst imaginable soreness

SECONDARY OUTCOMES:
Pressure pain threshold (PPT) of the hamstring muscles | change from before to after massage (average of 0, 10, 30 and 60 min after)
Hamstring range of motion | change from before to after massage (average of 0, 10, 30 and 60 min after)

CONTACTS AND LOCATIONS:
Overall Officials: Lars L Andersen, PhD, Principal Investigator — Professor
Locations (1):
- National Research Centre for the Working Environment, Copenhagen, Copenhagen, Denmark

REFERENCES:
- See also: Related Info — http://www.arbejdsmiljoforskning.dk